CLINICAL TRIAL: NCT06543992
Title: Efficacy and Safety of Intrathecal Administration of Thiotepa in Combination With Methotrexate Via the Ommaya Reservoir in Breast Cancer With Leptomeningeal Metastasis: a Phase II Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Intrathecal Administration of Thiotepa in Combination With Methotrexate in Breast Cancer With Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Brain Hospital of Nanjing Medical University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ommaya 01
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Leptomeningeal Metastasis of Breast Cancer
Keywords: methotrexate; thiotepa; intrathecal chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrathecal chemotherapy group (Experimental): Patients received intrathecal 15mg MTX combination with 10mg thiotepa twice a week for 2 weeks (4 injections) followed by monthly injections of 15mg MTX combination with 10mg thiotepa until an event that meets the criteria for termination occurs.
  Interventions: Drug: Intrathecal Administration of Thiotepa in Combination with Methotrexate via the Ommaya Reservoir

INTERVENTIONS:
Drug: Intrathecal Administration of Thiotepa in Combination with Methotrexate via the Ommaya Reservoir — Patients received intrathecal 15mg MTX combination with 10mg thiotepa twice a week for 2 weeks (4 injections) followed by monthly injections of 15mg MTX combination with 10mg thiotepa until an event that meets the criteria for termination occurs.

SUMMARY:
Evaluate the efficacy and safety of Intrathecal Administration of Thiotepa in Combination with Methotrexate via the Ommaya Reservoir in Breast Cancer with Leptomeningeal Metastasis

DETAILED DESCRIPTION:
This was a II, single-arm, prospective, multicenter study designed to estimate the efficacy and safety of intrathecal administration of thiotepa in combination with methotrexate via the Ommaya Reservoir in breast cancer with leptomeningeal metastasis.

The primary end point was iORR [complete response (CR) + partial response (PR)] according to RANO-LM. Scoring based on radiographic assessment in leptomeningeal metastases . A composite score (total score) is calculated and compared with the baseline total score. A 25% worsening in the current score relative to baseline defines radiographic progressive disease. A 50% improvement in the current score defines a radiographic partial response. Resolution of all baseline radiographic abnormalities defines a complete response. All other situations define stable disease. The secondary end points were changes in iPFS, iDoR, ORR, PFS, OS, DoR and exploratory analysis of the relationship between molecular markers and therapeutic efficacy.

This study is planned to include 22 patients with leptomeningeal metastasis from breast cancer who meet the entry criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult female ≥18 and ≤75 years old at the time of informed consent.
2. ECGO rating 0-3.
3. Histologically or cytologically confirmed breast cancer.
4. Cerebrospinal fluid cytology combined with central nervous system function and brain imaging demonstrated the diagnosis of breast cancer with meningeal metastases;
5. Patients can be implanted or have been implanted with Ommaya reservoirs;
6. Patient must have at least one measurable lesion (according to RECIST 1.1 criteria);
7. Postmenopausal or pre/perimenopausal female patients are eligible for enrolment; pre or perimenopausal female patients must be willing to receive LHRHa during the study period.
8. All patients were required to meet the following laboratory biochemical values prior to enrolment:

   * Haematology: Hb ≥90 g/L, WBC ≥3.5×109/L, ANC ≥1.5×109/L, PLT ≥100×109/L;
   * Liver function: for those without liver metastases, AST, ALT, ALP ≤2.5 times the upper limit of normal values, and ≤1.25 x the upper limit of normal values for total bilirubin; for those with liver metastases, AST, ALT, ALP ≤ 5 times the upper limit of normal value, and total bilirubin ≤ 1.5 x upper limit of normal value.

Exclusion Criteria:

1. Patients with other malignant tumors, excluding basal cell carcinoma and carcinoma in situ
2. Patients with severe or uncontrolled systemic disease, including uncontrolled hypertension or active bleeding tendency
3. The investigator considers the patient unsuitable for entry into this study.
4. Patients with toxicity from prior therapy that has not returned to normal or NCI-CTCAE grade 5.0
5. Patients who have a drug allergy or metabolic disorder to the drugs in this regimen
6. Pregnant or lactating women (women of childbearing age must have had a negative pregnancy test within 14 days prior to the first dose; if positive, pregnancy must be ruled out by ultrasound).
7. Patients who are concurrently enrolled in other clinical studies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Intracranial Overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Intracranial overall response rate (iORR) is defined as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR), as per local review and according to RANO-LM.

SECONDARY OUTCOMES:
Intracranial Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Intracranial progression-free survival (iPFS) is defined as the time from the date of randomization to the date of the first documented progression, as per local review and according to RANO-LM or death due to any cause.
Intracranial Duration of Response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Intracranial duration of response (iDoR) is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response, as per local review and according to RANO-LM.
Overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall response rate (ORR) is defined as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR), as per local review and according to RECIST 1.1.
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause.
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause
Duration of Response | From date of randomization until the date of death from any cause, assessed up to 100 months
  Duration of response (DoR) is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response, as per local review and according to RECIST 1.1.
frequency/severity of adverse events, lab abnormalities | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code